CLINICAL TRIAL: NCT05992090
Title: Neuromuscular Blockade Monitoring Using Kine-myography vs Electromyography in Patients Undergoing General Anaesthesia With the Use of Rocuronium and Cis-atracurium.
Brief Title: Neuromuscular Blockade Monitoring Using Kine-myography vs Electromyography.
Status: Completed | Type: Observational
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Michal Kalina, principal investigator, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Other Study IDs: EMG vs KMG
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Neuromuscular Blockade; Residual Neuromuscular Blockade
Keywords: neuromuscular blockade; electromyography; kine-myography; general anaesthesia; rocuronium; cis-atracurium; residual neuromuscular blockade; sugammadex
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare two monitoring methods of neuromuscular blockade - Kine-myography and Electromyography.

The main questions to answer are:

* are electromyography and kine-myography interchangeable
* is electromyography linked to fewer fault results
* is electromyography using lower energy to stimulate nerves

The type of study is a multicentric observational clinical trial. Subjects are patients undergoing general anaesthesia with the use of rocuronium or cis-atracurium. In each patient, the neuromuscular blockade will be monitored using kine-myograph and electromyography simultaneously.

DETAILED DESCRIPTION:
Informed consent will first be obtained from the patient for inclusion in the study. Consent will be obtained during an examination by the anaesthesiologist providing anaesthetic care during surgery in the anteroom of the operating theatre.

Once informed consent has been obtained, a routine orientation examination will be performed by the anaesthetist and routine pre-operative preparation (provision of peripheral venous access, risk assessment for airway obstruction, etc.) will be performed. The patient will then be transported to the operating theatre.

In the operating room, patient monitoring will be initiated, including the deployment of sensors to monitor the depth of neuromuscular blockade. The KMG sensor will be placed on the right arm and the EMG sensor on the left arm. After deployment of the sensors, upper limb fixation will be performed by the anaesthetic nurse. The fixation will be performed with splints compatible with the operating table. Fixation of the limbs and sensor with adhesive tape will not be used.

The anaesthesia will then be induced. Propofol and sufentanil will be administered at the discretion of the anaesthetist providing anaesthetic care. Once sufficient depth of sedation has been induced, calibration of the sensors monitoring the depth of neuromuscular blockade will be performed. After calibration of the sensors, the supramaximal current to the CRF will be recorded. The measurement interval will be set to 20 s. After securing the airway, the interval will be extended to 5 - 15 min according to the nature of the surgery and the discretion of the anaesthesiologist providing anaesthetic care. The number of twitches (PCT) and the Train Of Four (TOF) value will be recorded throughout the procedure.

On emergence from anaesthesia, the measurement interval will be set to 1 minute. Once sufficient depth of neuromuscular blockade has been reached to allow extubation, monitoring of the depth of neuromuscular blockade will be discontinued.

If during the measurement of the depth of neuromuscular blockade a value is measured that is highly suspected to be in error, this suspicion will be recorded in the CRF with a justification.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery under general anaesthesia with the use of cis-atracurium or rocuronium

Exclusion Criteria:

* patients suffering from neuromuscular diseases
* patients with known allergy to rocuronium or cis-atracurium
* patients in whom it is impossible to measure the depth of the neuromuscular block on the upper extremities (injuries of the upper extremities, contractures etc.)
* patients undergoing surgery positioned on their side
* patients with an upper arm injury
* patients with acromegaly
* patients with Alzheimer's disease
* patients with the risk of difficult airways
* patients induced into general anaesthesia via the Rapid Sequence Induction method
* patients with a weight under 5 kilograms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from residents of the Northern Bohemia region. All included patients will be indicated for surgery in general anesthesia with the need for neuromuscular blockade. All selected patients will be hospitalized at Masaryk Hospital in Ústí nad Labem.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Measurement variability | From sensor calibration til extubation at TOF higher than 90%.Maximum length of measurement is 6 hours.
  A primary aim is to demonstrate that measurement of the depth of neuromuscular blockade using kinemyography is associated with a higher measurement variability than measurement of the depth of neuromuscular blockade using electromyography.

SECONDARY OUTCOMES:
supramaximal electric stimulus | From sensor calibration til extubation at TOF higher than 90%.Maximum length of measurement is 6 hours.
  A secondary aim is to demonstrate that measuring the depth of neuromuscular blockade using kinemyography is associated with a higher supramaximal electric stimulus than measuring the depth of neuromuscular blockade using electromyography.
TOF overestimation | From sensor calibration til extubation at TOF higher than 90%.Maximum length of measurement is 6 hours.
  The primary objective of the study is to demonstrate that there is measured higher TOF when using KMG to monitor the depth of neuromuscular blockade compared to using EMG sensor to monitor the depth of neuromuscular blockade.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kalina, MUDr., Principal Investigator — Krajská Zdravotní a.s., Masarykova Nemocnice v Ústí nad Labem, Klinika anesteziologie, perioperační a intenzivní medicíny FZS UJEP a MNUL
Locations (1):
- Masarykova Nemocnice v Ústí nad Labem, Krajská Zdravotní a.s., Ústí nad Labem, Ústí Nad Labem Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided